CLINICAL TRIAL: NCT01157871
Title: Double-blind, Randomized, Placebo-controlled, Parallel Group and Dose-finding, Multicentric, Safety and Efficacy Study With Intramuscular Injections of NV1FGF in Subjects With Intermittent Claudication
Brief Title: Dose-finding, Safety and Efficacy Study of NV1FGF in Patients With Intermittent Claudication
Acronym: TALISMAN 211
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT6141; PM211 (Other: Gencell)
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Experimental): 4 administrations at 2-week interval of placebo solution
  Interventions: Drug: placebo
- NV1FGF 16 mg (Experimental): 4 administrations at 2-week interval of 4mg at each administration
  Interventions: Drug: XRP0038 (NV1FGF)
- NV1FGF 32 mg (Experimental): 4 administrations at 2-week interval of 8mg at each administration
  Interventions: Drug: XRP0038 (NV1FGF)

INTERVENTIONS:
Drug: XRP0038 (NV1FGF) — Pharmaceutical form:solution
  Route of administration: intramuscular
  Arms: NV1FGF 16 mg; NV1FGF 32 mg
Drug: placebo — Pharmaceutical form:solution
  Route of administration: intramuscular
  Arms: placebo

SUMMARY:
The primary objective is to assess safety and efficacy of two different doses of NV1FGF as compared to placebo.

The secondary objective is to assess the pharmacokinetics of NV1FGF and FGF-1 protein.

DETAILED DESCRIPTION:
Screening of 1 to 4 weeks before study drug administration; 6 weeks of treatment, followed by 20 weeks of follow-up.

ELIGIBILITY:
Inclusion criteria:

* Age>40 years
* History of typical intermittent claudication lasting for at least 3 months, showing no improvement and consistent with treadmill test findings
* Objective evidence of Peripheral Arterial Occlusive Disease. After 10 minutes of rest, either by Ankle brachial index measure (ABI) <0.8 or Systolic ankle pressure (AP) < 50 mmHg or Systolic toe pressure <50 mmHg
* Patent femoral inflow above the level of injections recently (<2 weeks) documented either with Doppler ultrasonography or Magnetic Resonance Angiography or Angiography

Exclusion criteria:

* Evidence of other causes for leg pain other than intermittent claudication.
* Illnesses limiting subject exercise capacity (angina pectoris, heart failure, respiratory disease, orthopaedic disease, neurological disorders…)
* Pain at rest
* Buerger's disease
* Positive serology for HIV 1 or 2, positive serology hepatitis B or C.
* Subjects with serum creatinine > 2 mg/dl (176 µmol/l) and subjects on dialysis.
* Active proliferative retinopathy defined by the presence of new vessel formation and scarring.
* Subjects who had a stroke or neurologic deficit presumed to be due to stroke within 3 months prior to the first administration of study treatment
* Previous treatment with any angiogenic growth factor
* Pregnant or breast feeding women or who disagree to practice a medically accepted method of birth control. Men and women who do not agree to use condoms as the only accepted protection barrier, for the entire study period
* Serious concomitant medical conditions not adequately controlled.
* Current alcohol or drug abuse

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Absolute Claudication Distance (ACD) evaluated by treadmill test at week 13 | 13 weeks

SECONDARY OUTCOMES:
NV1FGF DNA 69 base pair (bp) in plasma | up to week 27
NV1FGF DNA 825 bp in plasma | up to week 27
FGF-1 in plasma | up to week 27
Anti-FGF1 antibodies in serum | up to week 27

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Director — Sanofi
Locations (4):
- Minneapolis, Minnesota, United States
- Brussels, Belgium
- Münster, Germany
- Bern, Switzerland

REFERENCES:
- [Derived] Niebuhr A, Henry T, Goldman J, Baumgartner I, van Belle E, Gerss J, Hirsch AT, Nikol S. Long-term safety of intramuscular gene transfer of non-viral FGF1 for peripheral artery disease. Gene Ther. 2012 Mar;19(3):264-70. doi: 10.1038/gt.2011.85. Epub 2011 Jun 30. PMID 21716303